CLINICAL TRIAL: NCT06138938
Title: How Abdominal Irrigation During Cesarean Delivery Affects Gastrointestinal Functions and Short-term Maternal Morbidities: A Randomized Controlled Study
Brief Title: Effects of Abdominal Irrigation During Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Canan SATIR ÖZEL, MD, Gynecology and Obstetrics Specialist, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstanbulMU-CananSATIROZEL
Record Dates: First submitted 2023-09-15; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cesarean Section; Visual Analog Scale
Keywords: Abdominal irrigation; Cesarean section; Emesis; Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In the control group, abdominal irrigation as described in the study group was not performed.
- Study Group (Experimental): All blood clots and other remnants were manually externalized with a sponge holder forceps from the pelvic areas following the uterine incision closure. Then, 1,000 mL of warm saline irrigation was poured into the vesicouterine cavity and aspirated as much as possible in the reverse Trendelenburg position using an aspirator, carefully avoiding any contact with the intestines.
  Interventions: Other: Intraoperative abdominal irrigation

INTERVENTIONS:
Other: Intraoperative abdominal irrigation — All blood clots and other remnants were manually externalized with a sponge holder forceps from the pelvic areas following the uterine incision closure. Then, 1,000 mL of warm saline irrigation was poured into the vesicouterine cavity and aspirated as much as possible in the reverse Trendelenburg position using an aspirator, carefully avoiding any contact with the intestines.
  Arms: Study Group

SUMMARY:
This prospective randomized controlled clinical trial was conducted between March 2022 and May 2022 and included 60 patients who underwent elective cesarean. The participants were randomized into two groups: abdominal irrigation (n=30) and control group (n=30). Participants undergo a standard cesarean procedure, and general anesthesia was preferred. The patients were questioned regarding nausea, vomiting, highest pain scores, time of flatus, and stool passage during the postoperative period.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical study was conducted between March 2022 and May 2022. Ethical committee approval was obtained from the Istanbul Medeniyet University Göztepe Training and Research Hospital (decision no: 2022/0139, date: 16.03.2022). Informed consent was taken from each patient. The inclusion criteria for the study were term (≥37 weeks) and singleton pregnancies that underwent elective CS (cesarean section) under general anesthesia. The exclusion criteria were as follows: local anesthesia during surgery, chronic diseases including gastrointestinal, neurologic, and endocrinologic pathologies, CS with emergency indications, maternal coagulopathy, chorioamnionitis, placenta previa, placenta accreta, and mental retardation. Elective CS was defined as CS performed before the presence of labor with or without previous CS history. Primary CS was used for women without an earlier CS history.

All participants completed a questionnaire regarding their parity, age, body mass index, comorbidities, current medication, and tobacco use. Then, the patients were randomized into the control and study groups. The study group was composed of patients indicated for abdominal irrigation during CS. A random number table was used to assign patients to either one of the groups. Patients' treatments are held in sequentially numbered secure, opaque envelopes. After routine abdominal cleaning, surgeons were informed by the operating nurse, who opened the envelope for each randomized patient before the operation. A Foley catheter was inserted into every patient before CS. Povidone-iodine solution was used for skin preparation. General anesthesia was used for all participants. Patients indicated for regional anesthesia were excluded because they may experience nausea, even perioperatively; therefore, an additional antiemetic drug can affect the results. The first author and her team (obstetrics and gynecology surgeons: C.S.O. and Z.R.G) performed all procedures. Following Pfannenstiel incision, fascial aponeurosis was separated from the rectus abdominis muscles in cranial and caudal directions. The rectus muscles were divided on the midline after the caudal-cut aponeurosis was elevated under tension. The peritoneum was opened in an identical manner using a vertical midline incision. A bladder flap was not a routine step otherwise, if not necessary. Kerr incision was created with a scalpel, followed by blunt expansion. After the umbilical cord clamping, the anesthetist administered a 10 IU intravenous bolus of oxytocin over 5-10 second to each patient. The placenta was delivered. A total of 3,000 mL of lactated Ringer solution containing 60 IU of oxytocin was administered for 24 hour. Antibiotic prophylaxis with 1 g cefazolin was administered routinely, and no additional drugs were used during the operation. After the exteriorization of the uterus, the hysterotomy incision was closed.

All blood clots and other remnants were manually externalized with a sponge holder forceps from the pelvic areas following the uterine incision closure. Then, 1,000 mL of warm saline irrigation was poured into the vesicouterine cavity and aspirated as much as possible in the reverse Trendelenburg position using an aspirator, carefully avoiding any contact with the intestines.

The abdominal wall layers, including the peritoneum, were closed in every procedure. Subcutaneous tissue cauterization was performed to secure hemostasis. Moreover, 3-0 polyglactin 90 sutures were used to close the skin incision. Participants received the same postoperative care. Postoperative uterine contraction was checked every 15 minute for 2 hour and then every 4 hour. Urinary catheters were removed on the day after the operation. The physician staff responsible for collecting patients who reported nausea and vomiting symptoms was blinded to group randomization. Following the visual analog scale (VAS) explanation to all participants, the highest pain scores at 0-1, 4-6, 10-12, and 22-24 hour during postoperative follow-up were noted. On postoperative day 1, patients' surgical incisions were examined. Requirements for antiemetic drugs and return of gastrointestinal function were recorded, and a complete blood count was ordered for each patient. The primary outcome measured was the time of the first passage of flatus. Return of bowel function was defined as the passage of flatus. Secondary outcome measures were the occurrence of postoperative infections, including endometritis. On bimanual examination, postpartum endometritis was described as a body temperature over 38.5 °C in addition to the presence of foul-smelling discharge or unusually tender uterus. The body temperature should be ≥38 °C for at least 24 h after surgery, described as febrile morbidity, which was not related to other indications of infection. Wound infection was defined as the partial or total separation of the incision presenting with a purulent or serous wound discharge with induration, warmth, and tenderness.

To calculate intraoperative blood loss, the volume in the suction apparatus and used swabs were measured. After translating swab weights into mL, using blood density (1,050 g/mL), the irrigation amount (1,000 mL) was subtracted from the calculated volume.

Another researcher (H.N.D), who was blinded to the group assignments, recorded and analyzed the data.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were term (≥37 weeks) and singleton pregnancies that underwent elective CS (cesarean section) under general anesthesia.

Exclusion Criteria:

* The exclusion criteria were as follows: local anesthesia during surgery, chronic diseases including gastrointestinal, neurologic, and endocrinologic pathologies, CS with emergency indications, maternal coagulopathy, chorioamnionitis, placenta previa, placenta accreta, and mental retardation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 0-1, 4-6, 10-12, and 22-24 hour during postoperative follow-up
  The visual analog scale (VAS) explanation to all participants, the highest pain scores at 0-1, 4-6, 10-12, and 22-24 hour during postoperative follow-up were noted.
Gastrointestinal Functions | 0-48 hour during postoperative follow-up
  Time for passage of flatus (Return of bowel function was defined as the passage of flatus).

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Devrim Yardimci, Principal Investigator — Goztepe Prof Dr Süleyman Yalcin City Hospital; Abdulkadir Turgut, Study Chair — Istanbul Medeniyet University; Nisan Helin Donmez, Principal Investigator — Goztepe Prof Dr Süleyman Yalcin City Hospital; Zelal Rojda Gungordu, Principal Investigator — Goztepe Prof Dr Süleyman Yalcin City Hospital
Locations (1):
- Göztepe Prof Dr Süleyman Yalçın Şehir Hastanesi, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No